CLINICAL TRIAL: NCT00405860
Title: A Pilot Study of Mycophenolate Mofetil (MMF) in Patients With p-ANCA Microscopic Polyangiitis and Mild to Moderate Renal Dysfunction.
Brief Title: CellCept in p-ANCA Vasculitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Roche Pharma AG (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1679-02
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: MPO-ANCA Vasculitis; Microscopic Polyangiitis
MeSH Terms: conditions — Microscopic Polyangiitis | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: CellCept (mycophenolate mofetil)

SUMMARY:
Microscopic polyangiitis (MP) is a primary systemic vasculitis predominantly affecting small blood vessels. Following the widespread introduction of ANCA testing, the primary systemic vasculitis (SV), Wegener?s granulomatosis (WG) and microscopic polyangiitis (MP) appear to be more frequent than was previously thought (see definitions in Appendix 6). In addition, the existence of early and organ-limited forms of these diseases, such as renal-limited vasculitis (RLV) is now clearly recognized. Their annual incidence exceeds 20 per million per year and they account for at least 5 % of the causes of end stage renal failure. The two diseases share many features of their histology, serology and response to treatment, pointing to similarities in their pathogenesis, which have justified a common approach to their management. The standard treatment with corticosteroids (CS) and cyclophosphamide (CYC) is usually effective at controlling active disease but continued treatment is necessary to prevent disease relapse. Due to the cumulative toxicity associated with CYC treatment, alternatives have been looked for. Mycophenolate mofetil (MMF) has been used to treat patients with a variety of immune-mediated nephritides, including ANCA-associated vasculitis, with less toxicity than CYC but with variable outcome. The present trial will examine whether substitution of oral CYC with oral MMF is equally efficient for induction of remission with less adverse effects in cases of MP with mild to moderate renal involvement. All patients will receive the same regimen of oral prednisone + MMF. Prednisone will be tapered to a stop after 24 weeks but MMF will continue for a total of 18 months unless there is worsening or persistent disease. The trial ends after 18 months.

DETAILED DESCRIPTION:
1. Patients will receive I.V. methylprednisone, or I.V. dexamethazone, oral prednisone and oral MMF therapy as outlined in table 2.
2. MMF will be initiated within the first 1-2 weeks of the start of steroids. Patients will receive CellCept, 750 mg po b.i.d for the first week. Dose will be increased to 1000 mg po b.i.d for the second week, and thereafter, according to blood levels and patient tolerance. Target blood levels are 1 ? 3.5 g/ml. Treatment will be for a total of 18 months. This is based on the published dose-dependent adverse effect profiles in transplant patients (31-32) and on reports that lower doses are ineffective and shorter courses (less then 6 months) result in relapses or failure of therapy (25). Dose will be reduced in patient who can not tolerate MMF at the above dose.

2) Relapse treatment to follow guidelines for relapse regimens. 3) After 18 months, all medications will be tapered to a full stop unless disease is active or grumbling.

4) Pneumocystis pneumonia prophylaxis will be used during the trial (with sulfamethoxazole/trimethoprim, or Dapsone or Mepron if allergic to sulfa).

ELIGIBILITY:
1. Active microscopic polyangiitis
2. Active urinary sediment (>25 rbc/hpf, red cell casts or dysmorphic red cells)
3. Renal biopsy compatible with the diagnosis of microscopic polyangiitis, or diagnosis demonstrated by the presence of hematuria, proteinuria, and dysmorphic red blood cells, and / or red blood casts when biopsy is contraindicated.
4. Positive p-ANCA (MPO ELISA)
5. Serum creatinine < 3.0mg/dl.
6. Age 18 years or over.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is successful induction of remission as defined in Appendix 6 within 6 months.

SECONDARY OUTCOMES:
Major relapse necessitating a switch to induction OCS/CYC treatment or more aggressive treatment (e.g. plasma exchange).
Minor relapses that can effectively be controlled by a transient, non-toxic increase in OCS
Intolerance to trial medications and adverse effects. Adverse effects will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Silva F, Specks U, Kalra S, Hogan MC, Leung N, Sethi S, Fervenza FC. Mycophenolate mofetil for induction and maintenance of remission in microscopic polyangiitis with mild to moderate renal involvement--a prospective, open-label pilot trial. Clin J Am Soc Nephrol. 2010 Mar;5(3):445-53. doi: 10.2215/CJN.06010809. Epub 2010 Jan 21. PMID 20093349